CLINICAL TRIAL: NCT00224484
Title: A Study to Evaluate the Immunogenicity and Safety of GlaxoSmithKline Biologicals' Herpes Simplex Candidate Vaccine (gD2-AS04) in Healthy HSV Seronegative and Seropositive Female Subjects Aged 10-17 Years.
Brief Title: Safety Study of Herpes Simplex Vaccine in HSV Seronegative and Seropositive Females Between 10 and 17 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208141/040
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Herpes Simplex
Keywords: Herpes Simplex vaccine; Safety; Adolescents; Immunogenicity
MeSH Terms: conditions — Herpes Simplex | interventions — Herpes Simplex Virus Vaccines; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- GD2-AS04 GROUP (Experimental): Female subjects aged 10-17 years, who received 3 doses of gD2-AS04 vaccine, which were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
  Interventions: Biological: GSK208141
- HAVRIX GROUP (Active Comparator): Female subjects aged 10-17 years, who received 3 doses of Havrix, which were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
  Interventions: Biological: Havrix (investigational formulation)
- SALINE GROUP (Placebo Comparator): Female subjects aged 10-17 years, who received 3 doses of a saline solution, which were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GSK208141 — 3 intramuscular doses
  Other Names: Herpes simplex vaccine; gD2-AS04 vaccine
  Arms: GD2-AS04 GROUP
Biological: Havrix (investigational formulation) — 3 intramuscular doses
  Arms: HAVRIX GROUP
Biological: Placebo — 3 intramuscular doses
  Arms: SALINE GROUP

SUMMARY:
Main goal of this study is to compare the occurrence of serious adverse events (SAEs) between the herpes simplex (gD2-AS04) vaccine group and the Saline control group throughout the study period (up to month 12).

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Three groups of females (3000, 1500 and 1500 subjects, respectively) were injected 3 times (at months 0, 1 and 6) with the herpes simplex vaccine, the HavrixTM vaccine (control) and a Saline solution (placebo), respectively. Subjects were followed over 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that can and will comply with the requirements of the protocol should be enrolled in the study.
* Healthy female between, and including, 10 and 17 years of age at the time of the first vaccination.
* Written informed assent obtained from the subject and written informed consent obtained from a parent or legal guardian of the subject prior to enrolment. If the subject is above the legal age of consent in her country, written informed consent will only be obtained from the subject.
* Subjects must have a negative urine pregnancy test.
* Subjects of childbearing potential at the time of study entry must be abstinent or must be using an effective method of birth control for 30 days prior to vaccination and must agree to continue such precautions for two months after completion of the vaccination series. Subjects who reach menarche during the study and therefore are of childbearing potential must agree to follow the same precautions.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or likely to become pregnant during the first eight months of the study (months 0-8).
* Any previous confirmed history of, or current clinical signs or symptoms of, oro labial herpes (cold sores), herpetic whitlow or genital herpes disease, such as swelling, papules, vesicles, pustules, ulcers, crusts, fissures, erythema, discharge, dysuria or pain, burning, itching, tingling in the ano-genital area.
* History of previous or planned vaccination against hepatitis A or a history of hepatitis A infection.
* Previous vaccination against herpes.
* History of herpetic keratitis.
* History of multiform erythema.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of study vaccine with the following exceptions: administration of routine meningococcal, hepatitis B, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before and 30 days after the first dose of study vaccine.
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccines
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* History of a current acute or chronic autoimmune disease.
* History of any neurological disorders or seizures, with the exception of a single febrile seizure during childhood.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality
* Acute disease at the time of enrolment
* Oral temperature >= 37.5°C (99.5°F) / axillary temperature >= 37.5°C (99.5°F) at the time of enrolment.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5960 (Actual)
Dates: Start 2004-04-07 (Actual); Primary Completion 2007-07-24 (Actual); Study Completion 2007-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (129):
- United States (57):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Thornton, Colorado
  - GSK Investigational Site, Westminster, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa Beach, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Whitehouse Station, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Hilliard, Ohio
  - GSK Investigational Site, Pickerington, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Gray, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Magna, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Sandy City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Marshfield, Wisconsin
- Australia (5):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Carlton, Victoria
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Wilrijk
- Canada (6):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Beauport, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- GSK Investigational Site, Aarhus N, Denmark
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (15):
  - GSK Investigational Site, Château-Renault
  - GSK Investigational Site, Derval
  - GSK Investigational Site, Évreux
  - GSK Investigational Site, Haute-Goulaine
  - GSK Investigational Site, La Chapelle-sur-Erdre
  - GSK Investigational Site, Le Temple-de-Bretagne
  - GSK Investigational Site, Luynes
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nort-sur-Erdre
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pont-de-l'Arche
  - GSK Investigational Site, Saint-Aubin-des-Châteaux
  - GSK Investigational Site, Saint-Avertin
  - GSK Investigational Site, Saint-Sébastien-sur-Loire
  - GSK Investigational Site, Tours
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Komotini
  - GSK Investigational Site, Thessaloniki
- Hungary (6):
  - GSK Investigational Site, Bordány
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Hódmezővásárhely
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Zsombó
- Iceland (3):
  - GSK Investigational Site, Garðabaer
  - GSK Investigational Site, Kopavogur
  - GSK Investigational Site, Reykjavik
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Panevezys
  - GSK Investigational Site, Vilnius
- GSK Investigational Site, Rotterdam, Netherlands
- GSK Investigational Site, Christchurch, New Zealand
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
- GSK Investigational Site, Bucharest, Romania
- Spain (5):
  - GSK Investigational Site, Blanes
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Montgat/Barcelona
  - GSK Investigational Site, Valencia
- Sweden (6):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå
- United Kingdom (10):
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Bolton, Lancashire
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Coventry, West Midlands
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tavares F, Cheuvart B, Heineman T, Arellano F, Dubin G. Meta-analysis of pregnancy outcomes in pooled randomized trials on a prophylactic adjuvanted glycoprotein D subunit herpes simplex virus vaccine. Vaccine. 2013 Mar 25;31(13):1759-64. doi: 10.1016/j.vaccine.2013.01.002. Epub 2013 Jan 10. PMID 23313657
- [Background] HSV-040 Study Group; Abu-Elyazeed RR, Heineman T, Dubin G, Fourneau M, Leroux-Roels I, Leroux-Roels G, Richardus JH, Ostergaard L, Diez-Domingo J, Poder A, Van Damme P, Romanowski B, Blatter M, Silfverdal SA, Berglund J, Josefsson A, Cunningham AL, Flodmark CE, Tragiannidis A, Dobson S, Olafsson J, Puig-Barbera J, Mendez M, Barton S, Bernstein D, Mares J, Ratner P. Safety and immunogenicity of a glycoprotein D genital herpes vaccine in healthy girls 10-17 years of age: results from a randomised, controlled, double-blind trial. Vaccine. 2013 Dec 9;31(51):6136-43. doi: 10.1016/j.vaccine.2013.06.081. Epub 2013 Jul 9. PMID 23850416
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 208141/040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208141/040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208141/040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208141/040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208141/040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208141/040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Havrix Group: Female subjects aged 10-17 years, who received 3 doses of Havrix™, which were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
Period: Overall Study
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Started (5960 subjects were randomized, but only 5955 received vaccination) | 2977 | 1491 | 1487
Completed | 2831 | 1426 | 1425
Not Completed | 146 | 65 | 62
Not completed — Serious Adverse Event | 1 | 1 | 0
Not completed — Non-Serious Adverse Event | 5 | 7 | 3
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Withdrawal by Subject | 49 | 18 | 16
Not completed — Migrated/moved from study area | 18 | 5 | 5
Not completed — Lost to Follow-up | 66 | 28 | 36
Not completed — Reason not specified | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group | Total
Number analyzed (Participants) | 2977 | 1491 | 1487 | 5955
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.81 (2.21) | 13.81 (2.21) | 13.83 (2.21) | 13.81 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2977 | 1491 | 1487 | 5955
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 2650 | 1340 | 1330 | 5320
  Arabic/North African | 12 | 13 | 8 | 33
  East/South East Asian | 16 | 9 | 7 | 32
  South Asian | 6 | 2 | 6 | 14
  American Hispanic | 78 | 27 | 34 | 139
  Not specified | 58 | 22 | 31 | 111
  Black | 157 | 78 | 71 | 306

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 12
Population: The analyses were performed on the Total Vaccinated cohort, which included all subjects who received at least one dose of the study vaccine and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 2977 | 1491 | 1487
Participants | 71 | 42 | 37

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activities. Grade 3 redness/swelling = greater than (>) 30mm diameter and persisting more than 24 hours.
Time Frame: Within 7 days (Days 0-6) after each and any vaccination
Population: The analyses were performed on the Total Vaccinated cohort, only on subjects with their symptom sheets completed, who received at least one dose of the study vaccine and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 2970 | 1491 | 1484
Participants
  Pain, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Pain, Any, Dose 1 | 2120 | 508 | 247
  Pain, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Pain, Grade 3, Dose 1 | 106 | 9 | 6
  Redness, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Redness, Any, Dose 1 | 598 | 125 | 103
  Redness, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Redness, Grade 3, Dose 1 | 36 | 3 | 0
  Swelling, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Swelling, Any, Dose 1 | 464 | 66 | 50
  Swelling, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Swelling, Grade 3, Dose 1 | 36 | 1 | 5
  Pain, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1463
  Pain, Any, Dose 2 | 1685 | 389 | 189
  Pain, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1463
  Pain, Grade 3, Dose 2 | 90 | 9 | 4
  Redness, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1463
  Redness, Any, Dose 2 | 582 | 95 | 70
  Redness, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1463
  Redness, Grade 3, Dose 2 | 41 | 0 | 2
  Swelling, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1463
  Swelling, Any, Dose 2 | 499 | 38 | 31
  Swelling, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1463
  Swelling, Grade 3, Dose 2 | 49 | 0 | 3
  Pain, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Pain, Any, Dose 3 | 1729 | 377 | 161
  Pain, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Pain, Grade 3, Dose 3 | 137 | 12 | 2
  Redness, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Redness, Any, Dose 3 | 567 | 80 | 62
  Redness, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Redness, Grade 3, Dose 3 | 51 | 0 | 0
  Swelling, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Swelling, Any, Dose 3 | 540 | 46 | 32
  Swelling, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Swelling, Grade 3, Dose 3 | 47 | 0 | 3
  Pain, Any, Across doses | 2529 | 787 | 407
  Pain, Grade 3, Across doses | 278 | 26 | 12
  Redness, Any, Across doses | 1120 | 222 | 174
  Redness, Grade 3, Across doses | 107 | 3 | 2
  Swelling, Any, Across doses | 979 | 125 | 90
  Swelling, Grade 3, Across doses | 108 | 1 | 7

3. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, headache, malaise, rash, temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)] and urticaria. Any = occurrence of any general symptom regardless of intensity grade or relation to vaccination. Grade 3 arthralgia, fatigue, headache, malaise, rash = general symptom that prevented normal activity. Grade 3 temperature = greater than 39 degrees Celsius (°C). Grade 3 urticaria = urticaria distributed on at least 4 body areas. Related = general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 7 days (Days 0-6) after each and any vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 2970 | 1491 | 1484
Participants
  Arthralgia, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Arthralgia, Any, Dose 1 | 375 | 141 | 122
  Arthralgia, Related, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Arthralgia, Related, Dose 1 | 281 | 103 | 83
  Arthralgia, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Arthralgia, Grade 3, Dose 1 | 23 | 5 | 5
  Fatigue, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Fatigue, Any, Dose 1 | 864 | 377 | 384
  Fatigue, Related, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Fatigue, Related, Dose 1 | 603 | 246 | 247
  Fatigue, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Fatigue, Grade 3, Dose 1 | 51 | 24 | 17
  Headache, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Headache, Any, Dose 1 | 836 | 379 | 395
  Headache, Related, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Headache, Related, Dose 1 | 530 | 232 | 239
  Headache, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Headache, Grade 3, Dose 1 | 47 | 18 | 15
  Malaise, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Malaise, Any, Dose 1 | 515 | 213 | 225
  Malaise, Related, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Malaise, Related, Dose 1 | 354 | 138 | 146
  Malaise, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Malaise, Grade 3, Dose 1 | 48 | 18 | 13
  Rash, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Rash, Any, Dose 1 | 68 | 29 | 23
  Rash, Related, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Rash, Related, Dose 1 | 37 | 13 | 11
  Rash, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Rash, Grade 3, Dose 1 | 1 | 1 | 2
  Temperature (Orally), Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Temperature (Orally), Any, Dose 1 | 122 | 59 | 63
  Temperature(Orally), Related, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Temperature(Orally), Related, Dose 1 | 68 | 21 | 31
  Temperature(Orally), Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Temperature(Orally), Grade 3, Dose 1 | 6 | 5 | 4
  Urticaria, Any, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Urticaria, Any, Dose 1 | 27 | 10 | 16
  Urticaria, Related, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Urticaria, Related, Dose 1 | 18 | 3 | 10
  Urticaria, Grade 3, Dose 1: number analyzed (Participants) | 2966 | 1490 | 1482
  Urticaria, Grade 3, Dose 1 | 4 | 0 | 4
  Arthralgia, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Arthralgia, Any, Dose 2 | 259 | 102 | 54
  Arthralgia, Related, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Arthralgia, Related, Dose 2 | 219 | 77 | 39
  Arthralgia, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Arthralgia, Grade 3, Dose 2 | 24 | 6 | 2
  Fatigue, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Fatigue, Any, Dose 2 | 566 | 226 | 233
  Fatigue, Related, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Fatigue, Related, Dose 2 | 427 | 157 | 163
  Fatigue, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Fatigue, Grade 3, Dose 2 | 40 | 9 | 8
  Headache, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Headache, Any, Dose 2 | 579 | 282 | 245
  Headache, Related, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Headache, Related, Dose 2 | 387 | 192 | 157
  Headache, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Headache, Grade 3, Dose 2 | 44 | 15 | 7
  Malaise, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Malaise, Any, Dose 2 | 340 | 151 | 124
  Malaise, Related, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Malaise, Related, Dose 2 | 240 | 103 | 88
  Malaise, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Malaise, Grade 3, Dose 2 | 42 | 17 | 7
  Rash, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Rash, Any, Dose 2 | 57 | 16 | 20
  Rash, Related, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Rash, Related, Dose 2 | 39 | 10 | 17
  Rash, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Rash, Grade 3, Dose 2 | 2 | 1 | 1
  Temperature(Orally), Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Temperature(Orally), Any, Dose 2 | 126 | 58 | 55
  Temperature(Orally), Related, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Temperature(Orally), Related, Dose 2 | 63 | 17 | 27
  Temperature(Orally), Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Temperature(Orally), Grade 3, Dose 2 | 8 | 2 | 3
  Urticaria, Any, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Urticaria, Any, Dose 2 | 14 | 9 | 7
  Urticaria, Related, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Urticaria, Related, Dose 2 | 11 | 6 | 7
  Urticaria, Grade 3, Dose 2: number analyzed (Participants) | 2911 | 1466 | 1465
  Urticaria, Grade 3, Dose 2 | 1 | 1 | 1
  Arthralgia, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Arthralgia, Any, Dose 3 | 239 | 77 | 64
  Arthralgia, Related, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Arthralgia, Related, Dose 3 | 210 | 56 | 50
  Arthralgia, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Arthralgia, Grade 3, Dose 3 | 23 | 2 | 2
  Fatigue, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Fatigue, Any, Dose 3 | 539 | 213 | 201
  Fatigue, Related, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Fatigue, Related, Dose 3 | 429 | 158 | 143
  Fatigue, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Fatigue, Grade 3, Dose 3 | 32 | 13 | 15
  Headache, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Headache, Any, Dose 3 | 513 | 224 | 199
  Headache, Related, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Headache, Related, Dose 3 | 376 | 155 | 123
  Headache, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Headache, Grade 3, Dose 3 | 31 | 14 | 16
  Malaise, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Malaise, Any, Dose 3 | 321 | 112 | 118
  Malaise, Related, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Malaise, Related, Dose 3 | 248 | 77 | 81
  Malaise, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Malaise, Grade 3, Dose 3 | 39 | 10 | 15
  Rash, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Rash, Any, Dose 3 | 34 | 10 | 14
  Rash, Related, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Rash, Related, Dose 3 | 26 | 3 | 9
  Rash, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Rash, Grade 3, Dose 3 | 3 | 0 | 0
  Temperature (Orally), Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Temperature (Orally), Any, Dose 3 | 163 | 55 | 69
  Temperature(Orally), Related, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Temperature(Orally), Related, Dose 3 | 84 | 30 | 25
  Temperature(Orally), Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Temperature(Orally), Grade 3, Dose 3 | 11 | 1 | 3
  Urticaria, Any, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Urticaria, Any, Dose 3 | 16 | 10 | 6
  Urticaria, Related, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Urticaria, Related, Dose 3 | 11 | 7 | 5
  Urticaria, Grade 3, Dose 3: number analyzed (Participants) | 2852 | 1430 | 1435
  Urticaria, Grade 3, Dose 3 | 4 | 1 | 1
  Arthralgia, Any, Across doses | 585 | 233 | 192
  Arthralgia, Related, Across doses | 482 | 183 | 139
  Arthralgia, Grade 3, Across doses | 62 | 13 | 9
  Fatigue, Any, Across doses | 1176 | 524 | 526
  Fatigue, Related, Across doses | 913 | 382 | 376
  Fatigue, Grade 3, Across doses | 113 | 45 | 38
  Headache, Any, Across doses | 1240 | 579 | 549
  Headache, Related, Across doses | 875 | 408 | 364
  Headache, Grade 3, Across doses | 113 | 47 | 34
  Malaise, Any, Across doses | 834 | 362 | 347
  Malaise, Related, Across doses | 611 | 253 | 237
  Malaise, Grade 3, Across doses | 118 | 41 | 31
  Rash, Any, Across doses | 141 | 46 | 51
  Rash, Related, Across doses | 93 | 20 | 35
  Rash, Grade 3, Across doses | 6 | 2 | 3
  Temperature (Orally), Any, Across doses | 360 | 158 | 167
  Temperature (Orally), Related, Across doses | 193 | 65 | 77
  Temperature (Orally), Grade 3, Across doses | 23 | 8 | 10
  Urticaria, Any, Across doses | 50 | 25 | 27
  Urticaria, Related, Across doses | 37 | 15 | 21
  Urticaria, Grade 3, Across doses | 9 | 2 | 5

4. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 = event which prevented normal, everyday activities. In adults/ adolescents, such an AE would, for example, prevent attendance at work/ school and would necessitate the administration of corrective therapy. Related = event assessed by the investigator as causally related to study vaccination.
Time Frame: Within 30 days (Day 0-29) after any vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 2977 | 1491 | 1487
Participants
  Any AEs | 1325 | 676 | 667
  Grade 3 AEs | 154 | 68 | 83
  Related AEs | 313 | 136 | 128

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) With Medically Attended Visits
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. A medically attended visit is an event which prompted the subject to seek medical advice.
Time Frame: Within the 30 Day (Day 0-29) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 2977 | 1491 | 1487
Participants | 585 | 297 | 298

6. Secondary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCD)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: During the active phase (up to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 2977 | 1491 | 1487
Participants | 23 | 10 | 11

7. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed
Description: Assessed parameters were alanine aminotransferase (ALT), creatinine (CREA), haematocrit (Hct), platelets (PLA), red blood cells (RBC), urea and white blood cells (WBC). A subset of subjects was formed for these analyses. Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range at other timepoints. This outcome presents ALT results.
Time Frame: At months 7 and 12
Population: The analyses were performed on a subset of subjects from the Total Vaccinated cohort, which included subjects who received at least one dose of the study vaccine and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 530 | 257 | 273
Participants
  ALT, PRE NORMAL, M7- NORMAL: number analyzed (Participants) | 530 | 253 | 273
  ALT, PRE NORMAL, M7- NORMAL | 519 | 249 | 268
  ALT, PRE NORMAL, M7- BELOW: number analyzed (Participants) | 530 | 253 | 273
  ALT, PRE NORMAL, M7- BELOW | 2 | 1 | 0
  ALT, PRE NORMAL, M7- ABOVE: number analyzed (Participants) | 530 | 253 | 273
  ALT, PRE NORMAL, M7- ABOVE | 8 | 2 | 4
  ALT, PRE NORMAL, M7- MISSING: number analyzed (Participants) | 530 | 253 | 273
  ALT, PRE NORMAL, M7- MISSING | 1 | 1 | 1
  ALT, PRE NORMAL, M12- NORMAL: number analyzed (Participants) | 529 | 257 | 267
  ALT, PRE NORMAL, M12- NORMAL | 514 | 246 | 259
  ALT, PRE NORMAL, M12- BELOW: number analyzed (Participants) | 529 | 257 | 267
  ALT, PRE NORMAL, M12- BELOW | 4 | 1 | 2
  ALT, PRE NORMAL, M12- ABOVE: number analyzed (Participants) | 529 | 257 | 267
  ALT, PRE NORMAL, M12- ABOVE | 7 | 5 | 4
  ALT, PRE NORMAL, M12- MISSING: number analyzed (Participants) | 529 | 257 | 267
  ALT, PRE NORMAL, M12- MISSING | 4 | 5 | 2
  ALT, PRE BELOW, M7- NORMAL: number analyzed (Participants) | 4 | 4 | 4
  ALT, PRE BELOW, M7- NORMAL | 4 | 1 | 3
  ALT, PRE BELOW, M7- BELOW: number analyzed (Participants) | 4 | 4 | 4
  ALT, PRE BELOW, M7- BELOW | 0 | 3 | 1
  ALT, PRE BELOW, M7- ABOVE: number analyzed (Participants) | 4 | 4 | 4
  ALT, PRE BELOW, M7- ABOVE | 0 | 0 | 0
  ALT, PRE BELOW, M12- NORMAL: number analyzed (Participants) | 4 | 4 | 4
  ALT, PRE BELOW, M12- NORMAL | 4 | 2 | 3
  ALT, PRE BELOW, M12- BELOW: number analyzed (Participants) | 4 | 4 | 4
  ALT, PRE BELOW, M12- BELOW | 0 | 2 | 0
  ALT, PRE BELOW, M12- ABOVE: number analyzed (Participants) | 4 | 4 | 4
  ALT, PRE BELOW, M12- ABOVE | 0 | 0 | 0
  ALT, PRE BELOW, M12- MISSING: number analyzed (Participants) | 4 | 4 | 4
  ALT, PRE BELOW, M12- MISSING | 0 | 0 | 1
  ALT, PRE ABOVE, M7- NORMAL: number analyzed (Participants) | 11 | 10 | 7
  ALT, PRE ABOVE, M7- NORMAL | 4 | 5 | 2
  ALT, PRE ABOVE, M7- BELOW: number analyzed (Participants) | 11 | 10 | 7
  ALT, PRE ABOVE, M7- BELOW | 0 | 0 | 0
  ALT, PRE ABOVE, M7- ABOVE: number analyzed (Participants) | 11 | 10 | 7
  ALT, PRE ABOVE, M7- ABOVE | 3 | 2 | 3
  ALT, PRE ABOVE, M7- MISSING: number analyzed (Participants) | 11 | 10 | 7
  ALT, PRE ABOVE, M7- MISSING | 4 | 3 | 2
  ALT, PRE ABOVE, M12- NORMAL: number analyzed (Participants) | 12 | 9 | 7
  ALT, PRE ABOVE, M12- NORMAL | 4 | 5 | 1
  ALT, PRE ABOVE, M12- BELOW: number analyzed (Participants) | 12 | 9 | 7
  ALT, PRE ABOVE, M12- BELOW | 0 | 0 | 0
  ALT, PRE ABOVE, M12- ABOVE: number analyzed (Participants) | 12 | 9 | 7
  ALT, PRE ABOVE, M12- ABOVE | 5 | 3 | 3
  ALT, PRE ABOVE, M12- MISSING: number analyzed (Participants) | 12 | 9 | 7
  ALT, PRE ABOVE, M12- MISSING | 3 | 1 | 3

8. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed
Description: Assessed parameters were alanine aminotransferase (ALT), creatinine (CREA), haematocrit (Hct), platelets (PLA), red blood cells (RBC), urea and white blood cells (WBC). A subset of subjects was formed for these analyses. Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range at other timepoints. This outcome presents CREA results.
Time Frame: At months 7 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 586 | 282 | 300
Participants
  CREA, PRE NORMAL, M7- NORMAL | 543 | 268 | 284
  CREA, PRE NORMAL, M7- BELOW | 14 | 5 | 7
  CREA, PRE NORMAL, M7- ABOVE | 25 | 6 | 9
  CREA, PRE NORMAL, M7- MISSING | 4 | 3 | 0
  CREA, PRE NORMAL, M12- NORMAL: number analyzed (Participants) | 583 | 282 | 292
  CREA, PRE NORMAL, M12- NORMAL | 551 | 257 | 275
  CREA, PRE NORMAL, M12- BELOW: number analyzed (Participants) | 583 | 282 | 292
  CREA, PRE NORMAL, M12- BELOW | 11 | 7 | 6
  CREA, PRE NORMAL, M12- ABOVE: number analyzed (Participants) | 583 | 282 | 292
  CREA, PRE NORMAL, M12- ABOVE | 19 | 13 | 10
  CREA, PRE NORMAL, M12- MISSING: number analyzed (Participants) | 583 | 282 | 292
  CREA, PRE NORMAL, M12- MISSING | 2 | 5 | 1
  CREA, PRE BELOW, M7- NORMAL: number analyzed (Participants) | 43 | 23 | 15
  CREA, PRE BELOW, M7- NORMAL | 12 | 4 | 3
  CREA, PRE BELOW, M7- BELOW: number analyzed (Participants) | 43 | 23 | 15
  CREA, PRE BELOW, M7- BELOW | 31 | 19 | 10
  CREA, PRE BELOW, M7- ABOVE: number analyzed (Participants) | 43 | 23 | 15
  CREA, PRE BELOW, M7- ABOVE | 0 | 0 | 0
  CREA, PRE BELOW, M7- MISSING: number analyzed (Participants) | 43 | 23 | 15
  CREA, PRE BELOW, M7- MISSING | 0 | 0 | 2
  CREA, PRE BELOW, M12- NORMAL: number analyzed (Participants) | 41 | 22 | 14
  CREA, PRE BELOW, M12- NORMAL | 21 | 12 | 6
  CREA, PRE BELOW, M12- BELOW: number analyzed (Participants) | 41 | 22 | 14
  CREA, PRE BELOW, M12- BELOW | 20 | 10 | 8
  CREA, PRE BELOW, M12- ABOVE: number analyzed (Participants) | 41 | 22 | 14
  CREA, PRE BELOW, M12- ABOVE | 0 | 0 | 0
  CREA, PRE ABOVE, M7- NORMAL: number analyzed (Participants) | 37 | 20 | 23
  CREA, PRE ABOVE, M7- NORMAL | 15 | 4 | 11
  CREA, PRE ABOVE, M7- BELOW: number analyzed (Participants) | 37 | 20 | 23
  CREA, PRE ABOVE, M7- BELOW | 0 | 0 | 0
  CREA, PRE ABOVE, M7- ABOVE: number analyzed (Participants) | 37 | 20 | 23
  CREA, PRE ABOVE, M7- ABOVE | 22 | 16 | 12
  CREA, PRE ABOVE, M12- NORMAL: number analyzed (Participants) | 37 | 21 | 23
  CREA, PRE ABOVE, M12- NORMAL | 12 | 4 | 7
  CREA, PRE ABOVE, M12- BELOW: number analyzed (Participants) | 37 | 21 | 23
  CREA, PRE ABOVE, M12- BELOW | 0 | 0 | 0
  CREA, PRE ABOVE, M12- ABOVE: number analyzed (Participants) | 37 | 21 | 23
  CREA, PRE ABOVE, M12- ABOVE | 24 | 17 | 15
  CREA, PRE ABOVE, M12- MISSING: number analyzed (Participants) | 37 | 21 | 23
  CREA, PRE ABOVE, M12- MISSING | 1 | 0 | 1

9. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed
Description: Assessed parameters were alanine aminotransferase (ALT), creatinine (CREA), haematocrit (Hct), platelets (PLA), red blood cells (RBC), urea and white blood cells (WBC). A subset of subjects was formed for these analyses. Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range at other timepoints. This outcome presents Hct results.
Time Frame: At months 7 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 611 | 295 | 311
Participants
  Hct, PRE NORMAL, M7- NORMAL: number analyzed (Participants) | 611 | 294 | 311
  Hct, PRE NORMAL, M7- NORMAL | 562 | 279 | 287
  Hct, PRE NORMAL, M7- BELOW: number analyzed (Participants) | 611 | 294 | 311
  Hct, PRE NORMAL, M7- BELOW | 34 | 11 | 15
  Hct, PRE NORMAL, M7- ABOVE: number analyzed (Participants) | 611 | 294 | 311
  Hct, PRE NORMAL, M7- ABOVE | 8 | 2 | 3
  Hct, PRE NORMAL, M7- MISSING: number analyzed (Participants) | 611 | 294 | 311
  Hct, PRE NORMAL, M7- MISSING | 7 | 2 | 6
  Hct, PRE NORMAL, M12- NORMAL: number analyzed (Participants) | 607 | 295 | 303
  Hct, PRE NORMAL, M12- NORMAL | 562 | 275 | 276
  Hct, PRE NORMAL, M12- BELOW: number analyzed (Participants) | 607 | 295 | 303
  Hct, PRE NORMAL, M12- BELOW | 25 | 11 | 17
  Hct, PRE NORMAL, M12- ABOVE: number analyzed (Participants) | 607 | 295 | 303
  Hct, PRE NORMAL, M12- ABOVE | 12 | 2 | 3
  Hct, PRE NORMAL, M12- MISSING: number analyzed (Participants) | 607 | 295 | 303
  Hct, PRE NORMAL, M12- MISSING | 8 | 7 | 7
  Hct, PRE BELOW, M7- NORMAL: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M7- NORMAL | 20 | 8 | 10
  Hct, PRE BELOW, M7- BELOW: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M7- BELOW | 10 | 5 | 4
  Hct, PRE BELOW, M7- ABOVE: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M7- ABOVE | 0 | 0 | 0
  Hct, PRE BELOW, M7- MISSING: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M7- MISSING | 0 | 0 | 1
  Hct, PRE BELOW, M12- NORMAL: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M12- NORMAL | 17 | 9 | 9
  Hct, PRE BELOW, M12- BELOW: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M12- BELOW | 13 | 4 | 5
  Hct, PRE BELOW, M12- ABOVE: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M12- ABOVE | 0 | 0 | 0
  Hct, PRE BELOW, M12- MISSING: number analyzed (Participants) | 30 | 13 | 15
  Hct, PRE BELOW, M12- MISSING | 0 | 0 | 1
  Hct, PRE ABOVE, M7- NORMAL: number analyzed (Participants) | 14 | 11 | 10
  Hct, PRE ABOVE, M7- NORMAL | 11 | 8 | 8
  Hct, PRE ABOVE, M7- BELOW: number analyzed (Participants) | 14 | 11 | 10
  Hct, PRE ABOVE, M7- BELOW | 0 | 0 | 1
  Hct, PRE ABOVE, M7- ABOVE: number analyzed (Participants) | 14 | 11 | 10
  Hct, PRE ABOVE, M7- ABOVE | 3 | 2 | 1
  Hct, PRE ABOVE, M7- MISSING: number analyzed (Participants) | 14 | 11 | 10
  Hct, PRE ABOVE, M7- MISSING | 0 | 1 | 0
  Hct, PRE ABOVE, M12- NORMAL: number analyzed (Participants) | 14 | 10 | 9
  Hct, PRE ABOVE, M12- NORMAL | 11 | 8 | 9
  Hct, PRE ABOVE, M12- BELOW: number analyzed (Participants) | 14 | 10 | 9
  Hct, PRE ABOVE, M12- BELOW | 0 | 0 | 0
  Hct, PRE ABOVE, M12- ABOVE: number analyzed (Participants) | 14 | 10 | 9
  Hct, PRE ABOVE, M12- ABOVE | 2 | 2 | 0
  Hct, PRE ABOVE, M12- MISSING: number analyzed (Participants) | 14 | 10 | 9
  Hct, PRE ABOVE, M12- MISSING | 1 | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed
Description: Assessed parameters were alanine aminotransferase (ALT), creatinine (CREA), haematocrit (Hct), platelets (PLA), red blood cells (RBC), urea and white blood cells (WBC). A subset of subjects was formed for these analyses. Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range at other timepoints. This outcome presents PLA results.
Time Frame: At months 7 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 608 | 296 | 307
Participants
  PLA, PRE NORMAL, M7- NORMAL: number analyzed (Participants) | 608 | 294 | 307
  PLA, PRE NORMAL, M7- NORMAL | 576 | 286 | 292
  PLA, PRE NORMAL, M7- BELOW: number analyzed (Participants) | 608 | 294 | 307
  PLA, PRE NORMAL, M7- BELOW | 5 | 1 | 3
  PLA, PRE NORMAL, M7- ABOVE: number analyzed (Participants) | 608 | 294 | 307
  PLA, PRE NORMAL, M7- ABOVE | 20 | 4 | 5
  PLA, PRE NORMAL, M7- MISSING: number analyzed (Participants) | 608 | 294 | 307
  PLA, PRE NORMAL, M7- MISSING | 7 | 3 | 7
  PLA, PRE NORMAL, M12- NORMAL: number analyzed (Participants) | 603 | 296 | 299
  PLA, PRE NORMAL, M12- NORMAL | 579 | 278 | 284
  PLA, PRE NORMAL, M12- BELOW: number analyzed (Participants) | 603 | 296 | 299
  PLA, PRE NORMAL, M12- BELOW | 3 | 1 | 0
  PLA, PRE NORMAL, M12- ABOVE: number analyzed (Participants) | 603 | 296 | 299
  PLA, PRE NORMAL, M12- ABOVE | 12 | 9 | 5
  PLA, PRE NORMAL, M12- MISSING: number analyzed (Participants) | 603 | 296 | 299
  PLA, PRE NORMAL, M12- MISSING | 9 | 8 | 10
  PLA, PRE BELOW, M7- NORMAL: number analyzed (Participants) | 7 | 3 | 3
  PLA, PRE BELOW, M7- NORMAL | 2 | 1 | 1
  PLA, PRE BELOW, M7- BELOW: number analyzed (Participants) | 7 | 3 | 3
  PLA, PRE BELOW, M7- BELOW | 5 | 2 | 0
  PLA, PRE BELOW, M7- ABOVE: number analyzed (Participants) | 7 | 3 | 3
  PLA, PRE BELOW, M7- ABOVE | 0 | 0 | 1
  PLA, PRE BELOW, M7- MISSING: number analyzed (Participants) | 7 | 3 | 3
  PLA, PRE BELOW, M7- MISSING | 0 | 0 | 1
  PLA, PRE BELOW, M12- NORMAL: number analyzed (Participants) | 7 | 3 | 2
  PLA, PRE BELOW, M12- NORMAL | 2 | 2 | 1
  PLA, PRE BELOW, M12- BELOW: number analyzed (Participants) | 7 | 3 | 2
  PLA, PRE BELOW, M12- BELOW | 4 | 1 | 1
  PLA, PRE BELOW, M12- ABOVE: number analyzed (Participants) | 7 | 3 | 2
  PLA, PRE BELOW, M12- ABOVE | 0 | 0 | 0
  PLA, PRE BELOW, M12- MISSING: number analyzed (Participants) | 7 | 3 | 2
  PLA, PRE BELOW, M12- MISSING | 1 | 0 | 0
  PLA, PRE ABOVE, M7- NORMAL: number analyzed (Participants) | 35 | 19 | 25
  PLA, PRE ABOVE, M7- NORMAL | 29 | 11 | 14
  PLA, PRE ABOVE, M7- BELOW: number analyzed (Participants) | 35 | 19 | 25
  PLA, PRE ABOVE, M7- BELOW | 0 | 0 | 0
  PLA, PRE ABOVE, M7- ABOVE: number analyzed (Participants) | 35 | 19 | 25
  PLA, PRE ABOVE, M7- ABOVE | 6 | 8 | 11
  PLA, PRE ABOVE, M12- NORMAL: number analyzed (Participants) | 36 | 18 | 25
  PLA, PRE ABOVE, M12- NORMAL | 26 | 14 | 18
  PLA, PRE ABOVE, M12- BELOW: number analyzed (Participants) | 36 | 18 | 25
  PLA, PRE ABOVE, M12- BELOW | 0 | 0 | 0
  PLA, PRE ABOVE, M12- ABOVE: number analyzed (Participants) | 36 | 18 | 25
  PLA, PRE ABOVE, M12- ABOVE | 9 | 4 | 6
  PLA, PRE ABOVE, M12- MISSING: number analyzed (Participants) | 36 | 18 | 25
  PLA, PRE ABOVE, M12- MISSING | 1 | 0 | 1

11. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed
Description: Assessed parameters were alanine aminotransferase (ALT), creatinine (CREA), haematocrit (Hct), platelets (PLA), red blood cells (RBC), urea and white blood cells (WBC). A subset of subjects was formed for these analyses. Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range at other timepoints. This outcome presents RBC results.
Time Frame: At months 7 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 607 | 300 | 312
Participants
  RBC, PRE NORMAL, M7- NORMAL: number analyzed (Participants) | 607 | 298 | 312
  RBC, PRE NORMAL, M7- NORMAL | 580 | 284 | 295
  RBC, PRE NORMAL, M7- BELOW: number analyzed (Participants) | 607 | 298 | 312
  RBC, PRE NORMAL, M7- BELOW | 15 | 8 | 8
  RBC, PRE NORMAL, M7- ABOVE: number analyzed (Participants) | 607 | 298 | 312
  RBC, PRE NORMAL, M7- ABOVE | 6 | 3 | 2
  RBC, PRE NORMAL, M7- MISSING: number analyzed (Participants) | 607 | 298 | 312
  RBC, PRE NORMAL, M7- MISSING | 6 | 3 | 7
  RBC, PRE NORMAL, M12- NORMAL: number analyzed (Participants) | 603 | 300 | 305
  RBC, PRE NORMAL, M12- NORMAL | 574 | 281 | 280
  RBC, PRE NORMAL, M12- ABOVE: number analyzed (Participants) | 603 | 300 | 305
  RBC, PRE NORMAL, M12- ABOVE | 17 | 8 | 9
  RBC, PRE NORMAL, M12- BELOW: number analyzed (Participants) | 603 | 300 | 305
  RBC, PRE NORMAL, M12- BELOW | 5 | 4 | 9
  RBC, PRE NORMAL, M12- MISSING: number analyzed (Participants) | 603 | 300 | 305
  RBC, PRE NORMAL, M12- MISSING | 7 | 7 | 7
  RBC, PRE BELOW, M7- NORMAL: number analyzed (Participants) | 21 | 10 | 13
  RBC, PRE BELOW, M7- NORMAL | 10 | 8 | 7
  RBC, PRE BELOW, M7- BELOW: number analyzed (Participants) | 21 | 10 | 13
  RBC, PRE BELOW, M7- BELOW | 11 | 2 | 6
  RBC, PRE BELOW, M7- ABOVE: number analyzed (Participants) | 21 | 10 | 13
  RBC, PRE BELOW, M7- ABOVE | 0 | 0 | 0
  RBC, PRE BELOW, M12- NORMAL: number analyzed (Participants) | 21 | 10 | 13
  RBC, PRE BELOW, M12- NORMAL | 12 | 7 | 6
  RBC, PRE BELOW, M12- BELOW: number analyzed (Participants) | 21 | 10 | 13
  RBC, PRE BELOW, M12- BELOW | 9 | 3 | 7
  RBC, PRE BELOW, M12- ABOVE: number analyzed (Participants) | 21 | 10 | 13
  RBC, PRE BELOW, M12- ABOVE | 0 | 0 | 0
  RBC, PRE ABOVE, M7- NORMAL: number analyzed (Participants) | 26 | 10 | 11
  RBC, PRE ABOVE, M7- NORMAL | 19 | 7 | 7
  RBC, PRE ABOVE, M7- BELOW: number analyzed (Participants) | 26 | 10 | 11
  RBC, PRE ABOVE, M7- BELOW | 0 | 0 | 0
  RBC, PRE ABOVE, M7- ABOVE: number analyzed (Participants) | 26 | 10 | 11
  RBC, PRE ABOVE, M7- ABOVE | 5 | 2 | 4
  RBC, PRE ABOVE, M7- MISSING: number analyzed (Participants) | 26 | 10 | 11
  RBC, PRE ABOVE, M7- MISSING | 2 | 1 | 0
  RBC, PRE ABOVE, M12- NORMAL: number analyzed (Participants) | 26 | 8 | 9
  RBC, PRE ABOVE, M12- NORMAL | 17 | 5 | 7
  RBC, PRE ABOVE, M12- BELOW: number analyzed (Participants) | 26 | 8 | 9
  RBC, PRE ABOVE, M12- BELOW | 0 | 0 | 0
  RBC, PRE ABOVE, M12- ABOVE: number analyzed (Participants) | 26 | 8 | 9
  RBC, PRE ABOVE, M12- ABOVE | 7 | 3 | 1
  RBC, PRE ABOVE, M12- MISSING: number analyzed (Participants) | 26 | 8 | 9
  RBC, PRE ABOVE, M12- MISSING | 2 | 0 | 1

12. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed
Description: Assessed parameters were alanine aminotransferase (ALT), creatinine (CREA), haematocrit (Hct), platelets (PLA), red blood cells (RBC), urea and white blood cells (WBC). A subset of subjects was formed for these analyses. Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range at other timepoints. This outcome presents UREA results.
Time Frame: At months 7 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 651 | 310 | 329
Participants
  UREA, PRE NORMAL, M7- NORMAL | 632 | 304 | 316
  UREA, PRE NORMAL, M7- BELOW | 13 | 3 | 9
  UREA, PRE NORMAL, M7- ABOVE | 2 | 2 | 2
  UREA, PRE NORMAL, M7- MISSING | 4 | 1 | 2
  UREA, PRE NORMAL, M12- NORMAL: number analyzed (Participants) | 643 | 310 | 320
  UREA, PRE NORMAL, M12- NORMAL | 615 | 301 | 304
  UREA, PRE NORMAL, M12- BELOW: number analyzed (Participants) | 643 | 310 | 320
  UREA, PRE NORMAL, M12- BELOW | 18 | 5 | 10
  UREA, PRE NORMAL, M12- ABOVE: number analyzed (Participants) | 643 | 310 | 320
  UREA, PRE NORMAL, M12- ABOVE | 6 | 0 | 3
  UREA, PRE NORMAL, M12- MISSING: number analyzed (Participants) | 643 | 310 | 320
  UREA, PRE NORMAL, M12- MISSING | 4 | 4 | 3
  UREA, PRE BELOW, M7- NORMAL: number analyzed (Participants) | 9 | 10 | 9
  UREA, PRE BELOW, M7- NORMAL | 7 | 7 | 7
  UREA, PRE BELOW, M7- BELOW: number analyzed (Participants) | 9 | 10 | 9
  UREA, PRE BELOW, M7- BELOW | 2 | 3 | 2
  UREA, PRE BELOW, M7- ABOVE: number analyzed (Participants) | 9 | 10 | 9
  UREA, PRE BELOW, M7- ABOVE | 0 | 0 | 0
  UREA, PRE BELOW, M12- NORMAL: number analyzed (Participants) | 12 | 11 | 9
  UREA, PRE BELOW, M12- NORMAL | 10 | 6 | 8
  UREA, PRE BELOW, M12- BELOW: number analyzed (Participants) | 12 | 11 | 9
  UREA, PRE BELOW, M12- BELOW | 2 | 3 | 1
  UREA, PRE BELOW, M12- ABOVE: number analyzed (Participants) | 12 | 11 | 9
  UREA, PRE BELOW, M12- ABOVE | 0 | 0 | 0
  UREA, PRE BELOW, M12- MISSING: number analyzed (Participants) | 12 | 11 | 9
  UREA, PRE BELOW, M12- MISSING | 0 | 2 | 0
  UREA, PRE ABOVE, M7- NORMAL: number analyzed (Participants) | 5 | 4 | 1
  UREA, PRE ABOVE, M7- NORMAL | 3 | 3 | 0
  UREA, PRE ABOVE, M7- BELOW: number analyzed (Participants) | 5 | 4 | 1
  UREA, PRE ABOVE, M7- BELOW | 0 | 0 | 0
  UREA, PRE ABOVE, M7- ABOVE: number analyzed (Participants) | 5 | 4 | 1
  UREA, PRE ABOVE, M7- ABOVE | 2 | 1 | 1
  UREA, PRE ABOVE, M12- NORMAL: number analyzed (Participants) | 5 | 4 | 1
  UREA, PRE ABOVE, M12- NORMAL | 5 | 3 | 0
  UREA, PRE ABOVE, M12- BELOW: number analyzed (Participants) | 5 | 4 | 1
  UREA, PRE ABOVE, M12- BELOW | 0 | 0 | 0
  UREA, PRE ABOVE, M12- ABOVE: number analyzed (Participants) | 5 | 4 | 1
  UREA, PRE ABOVE, M12- ABOVE | 0 | 1 | 1

13. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed
Description: Assessed parameters were alanine aminotransferase (ALT), creatinine (CREA), haematocrit (Hct), platelets (PLA), red blood cells (RBC), urea and white blood cells (WBC). A subset of subjects was formed for these analyses. Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range at other timepoints. This outcome presents WBC results.
Time Frame: At months 7 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 579 | 274 | 286
Participants
  WBC, PRE NORMAL, M7- NORMAL: number analyzed (Participants) | 579 | 271 | 286
  WBC, PRE NORMAL, M7- NORMAL | 534 | 243 | 253
  WBC, PRE NORMAL, M7- BELOW: number analyzed (Participants) | 579 | 271 | 286
  WBC, PRE NORMAL, M7- BELOW | 34 | 23 | 17
  WBC, PRE NORMAL, M7- ABOVE: number analyzed (Participants) | 579 | 271 | 286
  WBC, PRE NORMAL, M7- ABOVE | 6 | 4 | 9
  WBC, PRE NORMAL, M7- MISSING: number analyzed (Participants) | 579 | 271 | 286
  WBC, PRE NORMAL, M7- MISSING | 5 | 1 | 7
  WBC, PRE NORMAL, M12- NORMAL: number analyzed (Participants) | 577 | 274 | 282
  WBC, PRE NORMAL, M12- NORMAL | 525 | 247 | 251
  WBC, PRE NORMAL, M12- BELOW: number analyzed (Participants) | 577 | 274 | 282
  WBC, PRE NORMAL, M12- BELOW | 31 | 13 | 17
  WBC, PRE NORMAL, M12- ABOVE: number analyzed (Participants) | 577 | 274 | 282
  WBC, PRE NORMAL, M12- ABOVE | 14 | 9 | 9
  WBC, PRE NORMAL, M12- MISSING: number analyzed (Participants) | 577 | 274 | 282
  WBC, PRE NORMAL, M12- MISSING | 7 | 5 | 5
  WBC, PRE BELOW, M7- NORMAL: number analyzed (Participants) | 64 | 35 | 36
  WBC, PRE BELOW, M7- NORMAL | 40 | 20 | 19
  WBC, PRE BELOW, M7- BELOW: number analyzed (Participants) | 64 | 35 | 36
  WBC, PRE BELOW, M7- BELOW | 22 | 13 | 17
  WBC, PRE BELOW, M7- ABOVE: number analyzed (Participants) | 64 | 35 | 36
  WBC, PRE BELOW, M7- ABOVE | 0 | 0 | 0
  WBC, PRE BELOW, M7- MISSING: number analyzed (Participants) | 64 | 35 | 36
  WBC, PRE BELOW, M7- MISSING | 2 | 2 | 0
  WBC, PRE BELOW, M12- NORMAL: number analyzed (Participants) | 62 | 32 | 31
  WBC, PRE BELOW, M12- NORMAL | 41 | 20 | 16
  WBC, PRE BELOW, M12- BELOW: number analyzed (Participants) | 62 | 32 | 31
  WBC, PRE BELOW, M12- BELOW | 20 | 10 | 12
  WBC, PRE BELOW, M12- ABOVE: number analyzed (Participants) | 62 | 32 | 31
  WBC, PRE BELOW, M12- ABOVE | 0 | 0 | 1
  WBC, PRE BELOW, M12- MISSING: number analyzed (Participants) | 62 | 32 | 31
  WBC, PRE BELOW, M12- MISSING | 1 | 2 | 2
  WBC, PRE ABOVE, M7- NORMAL: number analyzed (Participants) | 12 | 12 | 14
  WBC, PRE ABOVE, M7- NORMAL | 6 | 7 | 10
  WBC, PRE ABOVE, M7- BELOW: number analyzed (Participants) | 12 | 12 | 14
  WBC, PRE ABOVE, M7- BELOW | 0 | 0 | 0
  WBC, PRE ABOVE, M7- ABOVE: number analyzed (Participants) | 12 | 12 | 14
  WBC, PRE ABOVE, M7- ABOVE | 6 | 5 | 4
  WBC, PRE ABOVE, M12- NORMAL: number analyzed (Participants) | 12 | 12 | 14
  WBC, PRE ABOVE, M12- NORMAL | 4 | 9 | 11
  WBC, PRE ABOVE, M12- BELOW: number analyzed (Participants) | 12 | 12 | 14
  WBC, PRE ABOVE, M12- BELOW | 0 | 0 | 0
  WBC, PRE ABOVE, M12- ABOVE: number analyzed (Participants) | 12 | 12 | 14
  WBC, PRE ABOVE, M12- ABOVE | 8 | 3 | 3

14. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) With Medically Attended Visits
Description: as for outcome 5
Time Frame: Starting from Day 30 until the end of study (Month 18)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 2977 | 1491 | 1487
Participants | 397 | 201 | 188

15. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSC)
Description: MSCs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury. For outcomes covering the ESFU period, the Havrix Group and Saline Group were pooled.
Time Frame: During the Extended Safety Follow Up (ESFU) period (Month 12 to Month 18)
Population: The analyses were performed on the Total Vaccinated cohort, which included all subjects who received at least one dose of the study vaccine and for whom data were available. For the purpose of this analysis, the subjects from Havrix Group and Saline group were pooled into one group: Pooled Group.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Group: Pooled group of subjects 10-17 years of age from Havrix and Saline groups.
Arm/Group | gD2-AS04 Group | Pooled Group
Number analyzed (Participants) | 2977 | 2978
Participants | 69 | 73

16. Secondary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCD)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies. For outcomes covering the ESFU period, the Havrix Group and Saline Group were pooled.
Time Frame: During the Extended Safety Follow Up (ESFU) period (Month 12 to Month 18)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Pooled Group
Number analyzed (Participants) | 2977 | 2978
Participants | 1 | 0

17. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. For outcomes covering the ESFU period, the Havrix Group and Saline Group were pooled.
Time Frame: Up to month 18 (during active phase and ESFU period)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | gD2-AS04 Group | Pooled Group
Number analyzed (Participants) | 2977 | 2978
Participants | 90 | 100

18. Secondary Outcome: Anti-glycoprotein D (Anti-gD) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EU/mL). Analysis was based on an immunogenicity subset, stratified by initial serostatus: HSV seronegative (-)/ seropositive (+), this included gD2-AS04 vaccine recipients, as follows: HSV 1 and HSV 2 seronegative (HSV1-/2-) and HSV 1 seropositive and HSV 2 seronegative (HSV1+/2-)
Time Frame: At months 0, 7 and 12
Population: The analysis was performed on the ATP cohort for immunogenicity, in a predefined immunogenicity subset of HSV vaccine recipients (gD2-AS04 Group) who underwent assessment of biochemical and hematological parameters. Data from participants in the "Havrix Group" and "Saline Group" were not collected.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | gD2-AS04 Group
Number analyzed (Participants) | 386
EU/mL
  HSV1-2-, PRE: number analyzed (Participants) | 338
  HSV1-2-, PRE | 23.0 [21.7 to 24.4]
  HSV1-2-, M7 | 7808.6 [7185.3 to 8485.9]
  HSV1-2-, M12: number analyzed (Participants) | 380
  HSV1-2-, M12 | 2408.9 [2200.8 to 2636.7]
  HSV1+2-, PRE: number analyzed (Participants) | 190
  HSV1+2-, PRE | 1702.1 [1440.6 to 2011.0]
  HSV1+2-, M7: number analyzed (Participants) | 179
  HSV1+2-, M7 | 10344.1 [9552.2 to 11201.5]
  HSV1+2-, M12: number analyzed (Participants) | 170
  HSV1+2-, M12 | 6411.8 [5820.8 to 7062.9]

19. Secondary Outcome: Anti-deacylated Monophosphoryl Lipid A (Anti-MPL) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EU/mL). The subset of subjects used for this analysis was 50% of the pre-defined subset of subjects that underwent assessment of biochemical and hematological parameters.
Time Frame: At months 0, 7 and 12
Population: The analyses were performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects included in the immunogenicity subset for whom data concerning immunogenicity outcome measures were available (for whom assay results were available for antibodies against the study vaccine antigen component after Vaccination).
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | gD2-AS04 Group | Havrix Group | Saline Group
Number analyzed (Participants) | 303 | 128 | 151
EU/mL
  Anti-MPL, PRE: number analyzed (Participants) | 288 | 119 | 140
  Anti-MPL, PRE | 195.2 [172.6 to 220.8] | 168.3 [138.3 to 204.7] | 198.4 [166.4 to 236.5]
  Anti-MPL, M7 | 801.9 [722.7 to 889.7] | 152.7 [125.6 to 185.6] | 190.7 [159.7 to 227.7]
  Anti-MPL, M12: number analyzed (Participants) | 298 | 127 | 150
  Anti-MPL, M12 | 537.4 [488.9 to 590.8] | 193.8 [161.2 to 233.0] | 232.9 [198.3 to 273.5]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: -Group GD2-AS04, Group Havrix and Group Saline: during the active study period (Month 0 - 12). -GD2-AS04 (ESFU) Group and Pooled Group: during the combined active study period and the ESFU period (Month 0 - 18). Other Adverse Events: -Solicited local/general symptoms: during the 7-day post-vaccination period. -Unsolicited Adverse Events: during the 30-day post-vaccination.
Description: The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
  Other Adverse Events were not collected during the ESFU period, hence resulting in zero participants at risk for GD2-AS04 (ESFU) Group and Pooled Group.
Groups:
- Group GD2-AS04; GD2-AS04 (ESFU) Group: Female subjects aged 10-17 years, who received 3 doses of gD2-AS04 vaccine, which were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
- Group Havrix: Female subjects aged 10-17 years, who received 3 doses of Havrix™ vaccine, which were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
- Group Saline: Female subjects aged 10-17 years, who received 3 doses of a saline solution, which were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
- Pooled Group: Pooled group of subjects 10-17 years of age from Havrix and Saline groups, included in the Extended Safety Follow Up (ESFU) period.
Arm/Group | Group GD2-AS04 | Group Havrix | Group Saline | GD2-AS04 (ESFU) Group | Pooled Group
All-Cause Mortality (participants affected / at risk) | 0/2977 | 0/1491 | 0/1487 | 0/2977 | 0/2978
Serious Adverse Events (participants affected / at risk) | 71/2977 | 42/1491 | 37/1487 | 90/2977 | 100/2978
Other Adverse Events (participants affected / at risk) | 2718/2977 | 1210/1491 | 1082/1487 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group GD2-AS04 (N=2977) | Group Havrix (N=1491) | Group Saline (N=1487) | GD2-AS04 (ESFU) Group (N=2977) | Pooled Group (N=2978)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 1 | 0
Maculopathy (Eye disorders) | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Cyst (General disorders) | 0 | 1 | 0 | 0 | 1
Granuloma (General disorders) | 1 | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 9 | 3 | 3 | 11 | 8
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 2 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 2 | 0 | 1 | 3 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Peritonsillar abscess (Infections and infestations) | 2 | 1 | 0 | 2 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 2 | 0 | 1 | 2
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 1 | 3
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0 | 3
Tracheobronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Painful response to normal stimuli (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Peripheral nerve lesion (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 0 | 2 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 4 | 1 | 7
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Agression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Anorexia nervosa (Psychiatric disorders) | 1 | 1 | 1 | 1 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 2 | 2
Depression (Psychiatric disorders) | 6 | 0 | 2 | 8 | 5
Drug abuse (Psychiatric disorders) | 0 | 2 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 1 | 0 | 1 | 1
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 1 | 2 | 2
Suicide attempt (Psychiatric disorders) | 5 | 1 | 0 | 5 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0 | 1 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 2 | 1 | 0 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Encephalitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fusarium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Vertebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group GD2-AS04 (N=2977) | Group Havrix (N=1491) | Group Saline (N=1487) | GD2-AS04 (ESFU) Group (N=0) | Pooled Group (N=0)
Nasopharyngitis (Infections and infestations) | 147 | 75 | 81 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 151 | 50 | 69 | NA | NA
Pain (General disorders) | 2529/2970 | 787 | 407/1484 | NA | NA — The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Redness (General disorders) | 1120/2970 | 222 | 174/1484 | NA | NA — The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Swelling (General disorders) | 979/2970 | 125 | 90/1484 | NA | NA
Arthralgia (General disorders) | 585/2970 | 233 | 192/1484 | NA | NA — The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Fatigue (General disorders) | 1176/2970 | 524 | 526/1484 | NA | NA — The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Headache (General disorders) | 1240/2970 | 579 | 549/1484 | NA | NA — The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Malaise (General disorders) | 834/2970 | 362 | 347/1484 | NA | NA — The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Temperature (Orally) (General disorders) | 360/2970 | 158 | 167/1484 | NA | NA — The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.